CLINICAL TRIAL: NCT05580055
Title: Blood Donation of Healthy Blood for Prototype Testing at Entia
Brief Title: Blood Testing at Entia
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Entia Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 298186
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Healthy
MeSH Terms: interventions — Antibody Affinity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Capillary Sample: This group donates finger prick blood samples to Entia for the purpose of development.
  Interventions: Diagnostic Test: Affinity
- Venous Sample: This group donates venous blood samples to Enta, taken by a registered nurse.
  Interventions: Diagnostic Test: Affinity

INTERVENTIONS:
Diagnostic Test: Affinity — Blood Analyser

SUMMARY:
The investigators are recruiting healthy volunteers to donate a finger prick blood sample or a small venous sample to Entia for the further development and testing of our blood analyser. The venous samples are taken by a registered nurse hired via a third party company. The results of the blood tests are not informed to the participants unless they explicitly ask for it.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years and above
* healthy with no known conditions

Exclusion Criteria:

* Has a known health condition, including blood-borne diseases
* Inadequate understanding of the English language (written and verbal) that would require a translator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers, enrolled by invitation only
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-10-22 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
The difference in counts of the device tested blood vs the gold standard tested blood. | 3 years
  Venous blood drawn will be tested on a laboratory analyser, in which the results will be compared against the results when tested on Entia's analyser.

CONTACTS AND LOCATIONS:
Locations (1):
- Entia Ltd, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No